CLINICAL TRIAL: NCT02392221
Title: Impact of Therapeutic Strategies in the Pediatric Inflammatory Bowel Disease: a Population Based Study (1988-2011).
Acronym: Inspired
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Funding from DGOS (PHRC IR 2013 and PRME) (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI2013_843_0022
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Pediatric Inflammatory Bowel Disease
Keywords: Crohn's disease (CD); Pediatric; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Crohn's disease (CD) and ulcerative colitis (UC) are chronic Inflammatory Bowel Disease (IBD) and may affect all segments of the digestive tract.

DETAILED DESCRIPTION:
Crohn's disease (CD) and ulcerative colitis (UC) are chronic Inflammatory Bowel Disease (IBD) and may affect all segments of the digestive tract. These are diseases of multifactorial origin in which environmental and genetic factors are predominant.The EPIMAD registry, the world's largest epidemiological register for IBD, identifying all incident cases in the four departments of the North West of France showed between 1988 and 2007, an increase in the annual incidence of MC 71 % (6.5 / 105 (1988-1990) 11.1 / 105 (2006-2007) p <0.0001) in the age group 10-19 years. At the same time, the annual incidence of UC decreased 4.3 / 3.5 105 inhabitants / 105 inhabitants (20%), with phenotypic presentation remained stable. The increase in the incidence of CD will contribute to increase its weight in the health system, particularly in the pediatric CD frequently associated with an aggressive phenotype causing specific complications such as malnutrition, pubertal delay or thrive. These complications have a important impact on the quality of life with a long-term risk of functional disability. They may be associated with increased mortality. Immunosuppressants (azathioprine, methotrexate) have been used in pediatric forms only from the 90s and anti-TNF antibodies (infliximab and adalimumab), until the 2000s. These new therapeutic classes have profoundly changed the management of pediatric IBD. Although there is little data on the impact of these new treatments, early introduction of immunosuppressive and anti-TNFs seems to influence the natural history of IBD diagnosed in pediatric age. Anti-TNFs appear to be associated with more frequent and deeper remission. With the advent of these new treatment, new therapeutic targets such as endoscopic mucosal healing and more recently the deep remission combining clinical remission, biological and endoscopic, appears. However there is no data in the general population assessing the impact of new treatments and new therapeutic strategies in the pediatric population. Potential risks associated with the increasing use and early use of biological treatments in this particular population remain to be determined in the general population.

The main hypothesis of this study is that changes in therapeutic strategies in IBD diagnosed before 17 yeras old could influence the cumulative incidence of surgical resection and complications specific to this population as failure to thrive and delayed puberty, insertion socio-professional, the extension of the disease, hospitalization rates, and the rate of cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients in the pediatric cohort EPIMAD registry with a diagnosis of CD or UC or probable between 1988 and 2011.

Exclusion Criteria:

* None

Max Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric IBD patients in the area of EPIMAD registry Age of diagnosis < 17 years
Sampling Method: Non-Probability Sample
Enrollment: 966 (Actual)
Dates: Start 2015-05; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of surgical resection in CD and colectomy in pediatric UC | end of follow up
  Cumulative incidence of surgical resection in CD and colectomy in pediatric ulcerative colitis, depending on the date of diagnosis and the possibility of using immunosuppressants and / or anti-TNFs.

SECONDARY OUTCOMES:
Disease extension according to Montreal classification | end of follow up
  Phenotype of MICI maximum monitoring (Montreal classification), according to the date of diagnosis
Treatment during the follow up | end of follow up
  treatment
information about occurrence of postoperative complications | end of follow up
  Presence, date and type of occurrence of postoperative complications (Dindo classification).
Weight and size | end of follow up
  Weight and size at diagnosis, at the first intestinal resection and at the end of follow up
Hospitalisations | end of follow up
  number, duration, date
Studies category Socio-Professional | end of follow up
  Studies category Socio-Professional (CSP) and occupation
Age of puberty | end of follow up
  Age of puberty
Death | end of follow up
  Death and if so; due date and
Complications | end of follow up
  Serious infectious complications and cancer
cost-effectiveness evalutation of different management strategies of IBD | end of follow up
  cost-effectiveness evalutation of different management strategies of IBD according comparison of groups of patients
cost-effectiveness evalutation of different management strategies of IBD | end of follow up
  cost-effectiveness evalutation of different management strategies of IBD according the period of diagnosis
cost-effectiveness evalutation of different management strategies of IBD | end of follow up
  cost-effectiveness evalutation of different management strategies of IBD according Markov model of disease natural history
Variation of cost-effectiveness ratio of IBD treatment strategies | at 5 years
  Variation of cost-effectiveness ratio of IBD treatment strategies. Efficacy will be measured with number of avoided surgeries.
Variation of cost-effectiveness ratio of IBD treatment strategies | at 15 years
  Variation of cost-effectiveness ratio of IBD treatment strategies. Efficacy will be measured with number of avoided surgeries.
Variation of cost-utility ratio of IBD treatment strategies | at 15 years
  Variation of cost-utility ratio of IBD treatment strategies. Efficacy will be measured with number of avoided surgeries.

CONTACTS AND LOCATIONS:
Overall Officials: Mathurin Fumery, Doctor, Study Director — CHU Amiens France; Jean-Louis Dupas, professor, Study Director — CHU Amiens France
Locations (2):
- France (2):
  - CHRU Lille, Lille
  - CHU Rouen, Rouen